CLINICAL TRIAL: NCT02492880
Title: Study to Characterize the Effects of Programming Features of the Boston Scientific Precision Spectra™ Spinal Cord Stimulator System Using the CoverEdge™ Surgical Leads
Brief Title: CoverEdge Algorithm Programming Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 91051317
Record Dates: First submitted 2015-06-23; First posted 2015-07-09 (Estimated); Results first posted 2018-08-07 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Chronic Pain
Keywords: stimulation; implantable; pulse generator; back pain; chronic pain; leg pain
MeSH Terms: conditions — Chronic Pain; Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Precision Spectra™ SCS system programming features — Precision Spectra™ SCS system programming features using the CoverEdge surgical lead.

SUMMARY:
This is a prospective, on-label, multi-center, non-randomized, exploratory, single-arm study to characterize the effects of programming features of the Boston Scientific Precision Spectra™ Spinal Cord Stimulator (SCS) System using the CoverEdge™ surgical lead.

ELIGIBILITY:
Inclusion Criteria:

* Subject implanted, on-label, with a commercially approved Boston Scientific Spectra neurostimulation system and at least one CoverEdge or CoverEdge X surgical lead, per local directions for use (DFU).
* Subject signed a valid, Institutional Review Board (IRB)-approved informed consent form.
* Subject is 18 years of age or older when written informed consent is obtained.

Exclusion Criteria:

* Subject meets any contraindication in Boston Scientific (BSC) neurostimulation system local DFU.
* Subject is currently diagnosed with cognitive impairment, or exhibits any characteristic, that would limit study candidate's ability to assess pain relief or complete study assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-07-20 (Actual); Primary Completion 2017-02-21 (Actual); Study Completion 2017-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roshini Jain, Study Director — Boston Scientific Neuromodulation Corporation
Locations (2):
- United States (2):
  - Barolat Neuroscience, Denver, Colorado
  - Albany Medical Center, Albany, New York

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 15 subjects were enrolled in the study. 1 subject was enrolled in error who did not meet all inclusion criteria and was withdrawn and 1 subject was lost to follow-up prior to completing the Programming Visit. Statistically relevant conclusions cannot be made from this small sample size.
Period: Overall Study
Arm/Group | Precision Spectra™ SCS System Programming Features
Started | 15
Completed | 13
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Precision Spectra™ SCS System Programming Features
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Change in Paresthesia Distribution From Subject Completed Paresthesia Drawing Questionnaire
Description: Change in paresthesia distribution based on programming parameters
Time Frame: minimum 25 days post IPG implant
Measure: Count of Participants; unit: Participants
Arm/Group | Precision Spectra™ SCS System Programming Features
Number analyzed (Participants) | 13
Participants
  Yes | 13
  No | 0

ADVERSE EVENTS:
Arm/Group | Precision Spectra™ SCS System Programming Features
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-11): https://cdn.clinicaltrials.gov/large-docs/80/NCT02492880/Prot_SAP_000.pdf